CLINICAL TRIAL: NCT05828485
Title: A Single-dose, Open-label Clinical Study to Evaluate the Effect of Food on Pharmacokinetics of MY008211A Tablets in Healthy Adult Subjects
Brief Title: Effect of Food on Pharmacokinetics of MY008211A Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MY008211-1-03
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 : AB (Experimental): 6 subjects were given a single dose of MY008211A tablets in the fasting state and, after a 5-day washout period, a single dose of MY008211A tablet was administered after taking a standard high-fat and high-calorie fed.
  Interventions: Drug: MY008211A tablets
- Sequence 1 : BA (Experimental): 6 subjects were given a single dose of MY008211A tablet after taking a standard high-fat and high-calorie fed and, after a 5-day washout period, a single dose of MY008211A tablet in the fasting state.
  Interventions: Drug: MY008211A tablets

INTERVENTIONS:
Drug: MY008211A tablets — A single dose of MY008211A tablet was administered after fasting and high-fat, high-calorie feeding
  Other Names: no other name

SUMMARY:
This was a single-center, single-dose, open-label clinical study. 12 subjects were randomly assigned in a 1:1 ratio to one of the following dosing sequences (sequence 1: AB; Sequence 2: BA). Each dosing sequence consisted of two cycles, one dose per cycle, with a 5-day washout period between doses.

DETAILED DESCRIPTION:
A: A single dose of MY008211A tablets was administered in the fasting state (fasting for at least 10 h with water as needed).

B: A single dose of MY008211A tablets was administered after a standard high-fat, high-calorie fed.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age ≤ 45, male or female;
2. Body weight: ≥50 kg for male, ≥45 kg for female; body mass index (BMI): 19.0-26.0 kg/m2 (inclusive);
3. Informed consent will be signed before the trial, and the content, process and possible adverse reactions of the trial will be fully understood;
4. The volunteers should be able to communicate well with the researchers and understand and comply with the requirements of the study.

Exclusion Criteria:

1. Participants who were enrolled in a clinical trial or used a study drug within 3 months before administration of the study drug;
2. Patients with chronic or active gastrointestinal diseases such as esophageal disease, gastritis, gastric ulcer, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery within the past three years and still clinically relevant according to the investigator;
3. Patients with definite diseases of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, metabolic system and other diseases that require medical intervention or are not suitable for clinical trial (such as psychiatric history);
4. History of known or suspected immunodeficiency (e.g., history of frequent recurrent infections), inherited or acquired complement deficiency;
5. Patients had a clear history of capsular microbial infection within 6 months before screening; Including but not limited to: Streptococcus pneumoniae, Bacillus anthracis, Salmonella, Salmonella typhi, Klebsiella pneumoniae, Pseudomonas aeruginosa, Bacteroides fragilis, Neisseria meningitidis, Haemophilus influenzae, Legionella pneumophila infection history;
6. Patients with previous or current history of TB infection;
7. Active systemic bacterial, viral, or fungal infection within 14 days before administration of the study drug;
8. Fever (≥ 38 ° C) within 7 days before administration of the study drug;
9. Those who have a history of allergy to the trial preparation and any of its components or related preparations, or to drugs, foods or other substances;
10. Those who cannot tolerate intravenous puncture or have a history of syncope or needle sickness;
11. Patients who underwent surgery within 6 months before the study drug is used, which will be judged by the investigators to affect the absorption, distribution, metabolism, and excretion of the study drug; Surgical procedures within 4 weeks before the use of the study drug; Or planned to undergo a surgical procedure during the trial;
12. Who had taken any medicine (including Chinese herbal medicine, health products, etc.) within 14 days before administration of the study drug;
13. Who received a vaccine or live attenuated vaccine within 14 days before administration of the study drug, or who plan to receive a vaccine during the trial;
14. Who donated blood or lost a large amount of blood (> 400mL) within 3 months before administration of the study drug, received a blood transfusion or use of blood products, or intended to donate blood or blood components during or within 3 months after administration of the study drug;
15. Drug abusers or had used hard drugs (e.g., cocaine, phencyhexidine, etc.) or soft drugs (e.g., cannabis) within 1 year before administration of the study drug;
16. Smokers or had smoked more than 5 cigarettes per day in 3 months before study drug use, or will be unable to stop using any tobacco products during the study;
17. Heavy drinkers, who drink at least twice a day or more than 14 times a week, or are avid binge drinkers (one drink is defined as 125mL of wine, 220mL of beer, or 50mL of liquor; Binge drinking is defined as 5 or more drinks in approximately 2 hours); Or unwillingness to stop drinking alcohol or any alcohol-based product during the trial;
18. Those who have special requirements for diet and cannot abide by the uniform diet;
19. Volunteers (or their partners) who plan to be pregnant or donate sperm or eggs during the trial to 3 months after the end of the trial, or who are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, contraceptive rings, surgical sterilization, etc.);
20. Pregnant or lactating women; Or having unprotected sex within 2 weeks before using the study drug; Or oral contraceptive use within 30 days or long-acting estrogen or progestin injectable or implant use within 6 months before use of the study drug;
21. Physical examination, electrocardiogram, chest X-ray, abdominal ultrasound, vital signs, laboratory examination abnormalities were clinically significant (subject to clinician's judgment);
22. With positive uremic screening test;
23. With positive alcohol breath test;
24. Volunteers may not be able to complete the study for other reasons or have other reasons for not participating in the study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to 72 hours postdose
  Maximum Plasma Concentration (Cmax) Of MY008211A tablets
The Maximum Plasma Concentration (Tmax) | up to 72 hours postdose
  Time To Reach The Maximum Plasma Concentration (Tmax) Of MY008211A
Area Under The Concentration Versus Time Curve (AUC) | up to 72 hours postdose
  Area Under The Concentration Versus Time Curve (AUC) Of MY008211A

SECONDARY OUTCOMES:
The incidence and severity of adverse events to assess safety and tolerability | up to 9 days
  such as laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Wei feng, Ph.D, Study Chair — Wuhan Createrna Science and Technology Co., Ltd
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No